CLINICAL TRIAL: NCT00016289
Title: Phase II Study of Intraperitoneal Recombinant Human Interleukin-12 (rhIL-12) in Patients With Peritoneal Carcinomatosis (Residual Disease < 1cm) Associated With Ovarian Epithelial Cancer or Primary Peritoneal Carcinoma
Brief Title: Interleukin-12 in Treating Patients With Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02381; MDA-ID-00232; N01CM17003 (NIH); CDR0000068619 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Interleukin-12 Subunit p35; Interleukin-12

ARMS (1):
- Treatment (recombinant interleukin-12) (Experimental): Patients receive interleukin-12 intraperitoneally once weekly. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease receive 2 additional courses.
  Interventions: Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: recombinant interleukin-12 — Given intraperitoneally
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472

SUMMARY:
Phase II trial to study the effectiveness of intraperitoneal interleukin-12 in treating patients who have ovarian epithelial cancer or primary peritoneal cancer. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill tumor cells. Giving interleukin-12 directly into the peritoneal cavity may kill cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate and progression-free interval in patients with peritoneal carcinomatosis associated with ovarian epithelial cancer or primary peritoneal carcinoma treated with intraperitoneal interleukin-12.

II. Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients.

III. Determine peritoneal cavity tumor cell responses, in terms of negative cytology, conversion of aneuploidy to diploidy, and apoptosis as evidence of therapeutic effect, in patients treated with this regimen.

IV. Assess quality of life in patients treated with this regimen. V. Determine the pharmacology and pharmacokinetics of this drug in these patients.

VI. Determine whether this regimen facilitates adaptive or innate immunity in vivo or serum antibody responses to tumor-associated antigens in these patients.

VII. Determine whether this regimen decreases expression of vascular endothelial growth factor, fibroblast growth factor 2, and interleukin-8 as surrogate markers of angiogenesis and whether a decrease in marker expression is associated with clinical activity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive interleukin-12 intraperitoneally once weekly. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease receive 2 additional courses. Quality of life is assessed at baseline; prior to weeks 2, 4, 8, 12, and 16 of treatment; when patients are informed of their disease response; and then 2 weeks later. Patients are followed every 2 months for 1 year and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed peritoneal carcinomatosis associated with ovarian epithelial or primary peritoneal epithelial carcinoma

  * Surgically documented disease after prior platinum-based chemotherapy with or without surgery
  * Minimal residual disease, defined as metastases less than 1 cm in largest diameter
* No significant adhesions or symptoms of obstruction
* No extra-abdominal or parenchymal disease
* No more than 6 weeks since prior primary chemotherapy
* Performance status - Zubrod 0-1
* Absolute granulocyte count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Lymphocyte count greater than 600/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT no greater than 2.5 times upper limit of normal
* Albumin at least 3.0 g/dL
* Hepatitis B and C negative
* Creatinine no greater than 1.5 mg/dL
* No significant cardiac disease
* No significant pulmonary disease
* No overt autoimmune disease
* No other malignancy within the past 10 years except squamous cell carcinoma in situ or basal cell skin cancer
* HIV negative
* Successful placement of peritoneal catheter
* No prior immunotherapy
* See Disease Characteristics
* Recovered from prior chemotherapy
* No concurrent chemotherapy
* No chronic steroid therapy
* No prior radiotherapy
* See Disease Characteristics
* Recovered from prior surgery
* At least 2 weeks since prior laparoscopy
* At least 4 weeks since prior laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Rate of remission determined by laparoscopy or laparotomy | Up to 2 years
  Tested using an exact test for a single binomial proportion
Toxicity graded using the NCI CTC version 3.0 | Up to 2 years
  Evaluated for each dose level and each course of therapy.
Progression-free interval | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Renato Lenzi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States